CLINICAL TRIAL: NCT00150969
Title: Evaluation of the Clinical Use of Vitamin K Supplementation in Post-Menopausal Women With Osteopenia (ECKO Trial)
Brief Title: Vitamin K Supplementation in Post-Menopausal Osteopenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 01-0169; 50422 (Other Grant/Funding Number: Canadian Institute for Health Research (CIHR))
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Post-Menopausal Osteoporosis; Post-Menopausal Osteopenia
Keywords: vitamin K; bone mineral density; post-menopausal women; randomized double blind placebo controlled trial; osteoporosis; women's health
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — Vitamin K 1

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- phyloquinone (Experimental): 5 mg Vitamin K1
  Interventions: Dietary Supplement: vitamin K1 (phylloquinone)
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: vitamin K1 (phylloquinone)
  Arms: phyloquinone
Dietary Supplement: placebo — 1 pill daily
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether supplementation with 5 mg vitamin K daily over a 2-year period will prevent bone loss in post-menopausal women with osteopenia.

DETAILED DESCRIPTION:
Osteoporosis is major cause of morbidity and mortality in Canadian postmenopausal women. It is a systemic disease characterized by low bone mass and deterioration of bone microarchitecture, resulting in bone fragility and an increased risk of fractures. One in six women over the age of 50 have osteoporosis. The lifetime risk of an osteoporotic fracture for an average 50 year-old Canadian woman is >40%. The annual health care costs for osteoporotic fractures in Canada have been estimated to exceed $1.3 billion.

Recent data suggest that vitamin K supplements may decrease bone loss and prevent fractures. Vitamin K is a co-factor of gamma-glutamyl carboxylase, an enzyme that catalyzes the gamma-carboxylation of glutamic acid residues in bone matrix proteins such as osteocalcin. Vitamin K has been reported to enhance bone formation in both in vitro studies and in vivo studies in animals. Vitamin K levels are low in individuals with osteoporosis and in patients with osteoporotic fractures. The few studies examining vitamin K supplementation in humans have showed promising results with no significant side effects, but these studies had significant methodological shortcomings such as inadequate sample size and lack of randomization.

The primary objective of our study is to examine whether vitamin K supplementation will increase bone mineral density in postmenopausal women with osteopenia. Our secondary objectives are to examine the possible adverse effects from long-term vitamin K supplementation, to investigate whether vitamin K will decrease risk of fractures and to determine if vitamin K affects quality of life. Our hypotheses are that vitamin K increases bone mineral density in postmenopausal women, and that there are no significant adverse effects from vitamin K supplementation.

ELIGIBILITY:
Inclusion Criteria:

Postmenopausal: One year since the natural cessation of menses, or Hysterectomy with either postmenopausal status confirmed by FSH lab values, or age 55 and above AND 2. Osteopenic: T-score at baseline has to be between (and including) -1.0 and

-2.0 in the lumbar spine (L1-L4), total hip or femoral neck, and the lowest reading of the above three measurements must be between -1.0 and -2.0

Exclusion Criteria:

1. Women ever having had a fragility fracture after age 40;
2. Women currently on anticoagulants, previously on anticoagulants in the past 3 months, or expected to be on anticoagulants in the near future;
3. Women on hormone replacement therapy, raloxifene, bisphosphonates or calcitonin during the past 3 months;
4. Women who have ever been on a bisphosphonate for more than 6 months;
5. Women previously diagnosed with Paget's disease, hyperparathyroidism, hyperthyroidism or other metabolic bone diseases;
6. Women with decompensated diseases of the liver, kidney, pancreas, lung, or heart;
7. Women with a history of active cancer in the past 5 years;
8. Women taking mega-doses of vitamin A (more than 10,000 iu per day) or E (more than 400 iu per day);
9. Women involved in other clinical trials;
10. Any women who, in the opinion of the principal investigator, is at poor medical or psychiatric risk for the study.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2002-01; Primary Completion 2006-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela M Cheung, MD, PhD, Principal Investigator — University Health Network, University of Toronto
Locations (5):
- Canada (5):
  - St. Michael's Hospital Health Centre, Toronto, Ontario
  - Mt. Sinai Hospital, Toronto, Ontario
  - University Health Network, Osteoporosis Department, Toronto, Ontario
  - Sunnybrook & Women's College Health Sciences Centre, Toronto, Ontario
  - University of Toronto, Toronto, Ontario

REFERENCES:
- [Result] Cheung AM, Tile L, Lee Y, Tomlinson G, Hawker G, Scher J, Hu H, Vieth R, Thompson L, Jamal S, Josse R. Vitamin K supplementation in postmenopausal women with osteopenia (ECKO trial): a randomized controlled trial. PLoS Med. 2008 Oct 14;5(10):e196. doi: 10.1371/journal.pmed.0050196. PMID 18922041

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment from January 2002 to September 2006 through health fairs, community posters and advertisements.
Pre-assignment Details: 453 participants signed consent. 13 were not included in analysis(10 screen failure,3 drop out at baseline)
Groups:
- Placebo: dummy pill identicle to vitamin k
Period: 24 Month Main Study
Arm/Group | Phyloquinone | Placebo
Started | 217 | 223
Completed | 198 | 202
Not Completed | 19 | 21
Not completed — Adverse Event | 3 | 4
Not completed — Death | 1 | 1
Not completed — Lack of Efficacy | 1 | 8
Not completed — Lost to Follow-up | 3 | 2
Not completed — Protocol Violation | 4 | 2
Not completed — Withdrawal by Subject | 7 | 4
Period: 24-48 Month Extension
Arm/Group | Phyloquinone | Placebo
Started | 121 | 140
Completed | 33 | 40
Not Completed | 88 | 100
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Lack of Efficacy | 0 | 1
Not completed — Adverse Event | 1 | 3
Not completed — Other Reason | 81 | 91

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phyloquinone | Placebo | Total
Number analyzed (Participants) | 217 | 223 | 440
Age, Continuous [Mean (Full Range); unit: years] | 58.9 [40.1 to 80.5] | 59.2 [46.1 to 82.3] | 59.0 [40.1 to 82.3]
Sex: Female, Male [Count of Participants; unit: Participants] — All Participants were community dwelling post-menopausal women
  Participants
    Female | 217 | 223 | 440
    Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Bone Mineral Density (BMD) at the Lumbar Spine (L1-L4) Between Treatment Arms.
Description: BMD was measured yearly on one scanner at UHN using DEXA Hologic 4500A densitometer
Time Frame: 0 to 24 months
Population: For our 2 year BMD anlayses we included all 440 women based on intention to treat using last observation carried forward for missing data.
Measure: Mean (Standard Deviation); unit: percentage change in BMD
Groups:
- Phyloquinone: 5 mg Vitamin K1 daily
Arm/Group | Phyloquinone | Placebo
Number analyzed (Participants) | 217 | 223
percentage change in BMD | -1.28 (3.5) [-0.67 to 0.54] | -1.22 (3.0) [-0.67 to 0.54]
Statistical Analysis 1: Comparison: Phyloquinone vs Placebo; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

2. Secondary Outcome: Percent Change in Bone Mineral Density (BMD) at the Femoral Neck Between Treatment Arms.
Description: BMD was measured yearly on one scanner at UHN using DEXA Hologic 4500A densitometer
Time Frame: 0 to 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage change in BMD
Arm/Group | Phyloquinone | Placebo
Number analyzed (Participants) | 217 | 223
percentage change in BMD | -1.47 (3.7) | -1.83 (3.5)

3. Secondary Outcome: Percent Change in Bone Mineral Density (BMD) at the Ultra-distal Radius Between Treatment Arms.
Description: BMD was measured yearly on one scanner at UHN using DEXA Hologic 4500A densitometer
Time Frame: 0 to 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage change in BMD
Arm/Group | Phyloquinone | Placebo
Number analyzed (Participants) | 217 | 221
percentage change in BMD | -2.49 (4.0) | -2.55 (4.7)

4. Secondary Outcome: Effect of Vitamin K1 Supplementation on Levels of Bone Formation Marker
Description: measured by osteocalcin on elecsys platform
Time Frame: 0-24 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Phyloquinone | Placebo
Number analyzed (Participants) | 198 | 192
ng/ml | 21 (7.3) | 24 (7.5)

5. Secondary Outcome: Effect of Vitamin K1 Supplementation on Level of Bone Resorption Markers (C-telopeptide: CTX)
Description: measured by CTX Elisa assay on elecsys platform
Time Frame: 0-24 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Phyloquinone | Placebo
Number analyzed (Participants) | 192 | 198
ng/ml | 0.58 (0.21) | 0.54 (0.21)

6. Secondary Outcome: Effect of Vitamin K1 Supplementation on Percent of Carboxylation of Osteocalcin
Description: measured by osteocalcin hydroxyapatite binding assay
Time Frame: 0 to 24 months
Measure: Mean (Standard Deviation); unit: percentage of undercarboxylated OC
Arm/Group | Phyloquinone | Placebo
Number analyzed (Participants) | 192 | 198
percentage of undercarboxylated OC | -21.4 (10.3) | -2.0 (6.8)

7. Secondary Outcome: Percent Change in Bone Mineral Density (BMD) at the Total Hip Between Treatment Arms.
Description: BMD was measured yearly on one scanner at UHN using DEXA Hologic 4500A densitometer
Time Frame: 0 to 48 months
Measure: Mean (Standard Deviation); unit: percentage change in BMD
Arm/Group | Phyloquinone | Placebo
Number analyzed (Participants) | 33 | 40
percentage change in BMD | -1.39 (3.6) | -1.52 (4.5)

8. Primary Outcome: Percent Change in Bone Mineral Density (BMD) at the Total Hip Between Treatment Arms.
Description: BMD was measured yearly on one scanner at UHN using DEXA Hologic 4500A densitometer
Time Frame: 0 to 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage change in BMD
Arm/Group | Phyloquinone | Placebo
Number analyzed (Participants) | 217 | 223
percentage change in BMD | -0.69 (2.8) [-0.37 to 0.75] | -0.88 (3.2) [-0.37 to 0.75]
Statistical Analysis 1: Comparison: Phyloquinone vs Placebo; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

9. Secondary Outcome: Percent Change in Bone Mineral Density (BMD) at the Lumbar Spine (L1-L4) Between Treatment Arms.
Description: BMD was measured yearly on one scanner at UHN using DEXA Hologic 4500A densitometer
Time Frame: 0 to 48 months
Measure: Mean (Standard Deviation); unit: percentage change in BMD
Arm/Group | Phyloquinone | Placebo
Number analyzed (Participants) | 33 | 40
percentage change in BMD | -0.40 (4.7) | -1.76 (3.8)

10. Secondary Outcome: Percent Change in Bone Mineral Density (BMD) at the Femoral Neck Between Treatment Arms.
Description: BMD was measured yearly on one scanner at UHN using DEXA Hologic 4500A densitometer
Time Frame: 0 to 48 months
Measure: Mean (Standard Deviation); unit: percentage change in BMD
Arm/Group | Phyloquinone | Placebo
Number analyzed (Participants) | 33 | 40
percentage change in BMD | -2.05 (4.3) | -2.71 (4.8)

11. Secondary Outcome: Percent Change in Bone Mineral Density (BMD) at the Ultra-distal Radius Between Treatment Arms.
Description: BMD was measured yearly on one scanner at UHN using DEXA Hologic 4500A densitometer
Time Frame: 0 to 48 months
Measure: Mean (Standard Deviation); unit: percentage change in BMD
Arm/Group | Phyloquinone | Placebo
Number analyzed (Participants) | 33 | 40
percentage change in BMD | -5.35 (5.1) | -5.23 (4.5)

12. Secondary Outcome: Difference in Serious Adverse Events
Description: These include hospitalizations for pneumonia, heart failure, gastro-intestinal bleeding, elective and non-elective surgery, cancer and death.
Time Frame: up to 48 months
Measure: Number; unit: events
Arm/Group | Phyloquinone | Placebo
Number analyzed (Participants) | 217 | 223
events | 15 | 25

13. Secondary Outcome: Difference in Number of New Cancers by Treatment Arm.
Time Frame: up to 48 months
Measure: Number; unit: events
Arm/Group | Phyloquinone | Placebo
Number analyzed (Participants) | 217 | 223
events | 3 | 12

14. Secondary Outcome: Difference in Number of New Clinical Fractures by Treatment Arm.
Description: these included fragility fractures
Time Frame: up to 48 months
Measure: Number; unit: events
Arm/Group | Phyloquinone | Placebo
Number analyzed (Participants) | 217 | 223
events | 11 | 21

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the entire study period of 48 months
Arm/Group | Phyloquinone | Placebo
Serious Adverse Events (participants affected / at risk) | 15/217 | 25/223
Other Adverse Events (participants affected / at risk) | 11/217 | 10/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phyloquinone (N=217) | Placebo (N=223)
hospitalization (General disorders) | 11 (13) | 13 (16) — these include pneumonia, heart failure, gastro-intestinal bleeding, elective and non-elective surgeries.
Cancer (General disorders) | 3 (3) | 11 (12) — cancers include uterine (2), vaginal(1), esophagus(1), thyroid(3), breast(7), lung (1)
Death (General disorders) | 1 (1) | 1 (4) — Causes of death include motor vehicle accident (1), arrhthmogenic right ventricular cardiomyopathy(1) cancer(3),
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phyloquinone (N=217) | Placebo (N=223)
nausea and vomitting (Gastrointestinal disorders) | 11 (11) | 10 (10)

LIMITATIONS AND CAVEATS:
Originally designed as a 2-year study with BMD as primary outcome. Thus, the number of women followed to 3 and 4 years was small, and the study was not powered to examine fracture outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes